CLINICAL TRIAL: NCT05782972
Title: Therapeutic Response of Sodium-glucose Co-transporter Type-2 Inhibitor in Non-diabetic MAFLD Patients: a Pilot Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Chia-Chi Wang, Professor, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCRD-TPE-112-11
Record Dates: First submitted 2023-02-19; First posted 2023-03-24 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Metabolic Associated Fatty Liver Disease
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: single-arm, prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- dapagliflozin (Forxiga) treatment (Experimental): The participants received oral dapagliflozin (Forxiga) 10 mg/day for 24 weeks
  Interventions: Drug: dapagliflozin (Forxiga)

INTERVENTIONS:
Drug: dapagliflozin (Forxiga) — The participants received oral dapagliflozin (Forxiga) 10 mg/day for 24 weeks.

SUMMARY:
The goal of this single arm, prospective study is to test the therapeutic response of oral dapagliflozin (Forxiga) 10 mg/day for 24 weeks in non-diabetic MAFLD patients. The primary outcomes are the improvement of liver inflammation or fibrosis parameters after 24 weeks treatment. The adverse events were also recorded.

DETAILED DESCRIPTION:
This is single-arm, prospective study and 50 non-diabetic MAFLD patients are enrolled consecutively at Taipei Tzu Chi Hospital. The non-diabetic definition is no previous history of diabetes mellitus and HbA1C < 6.5%. Fatty liver was diagnosed by imaging such as liver ultrasound or histologic examination. Metabolic dysfunction was defined as overweight/obese, or more than 2 metabolic abnormalities in lean/normal weight subjects. Inclusion criteria were ALT elevation (>35 U/L in male and >25 U/L in female) or FIB-4 >=1.45. Those with cancer history, systolic blood pressure < 100 mmHg, or eGFR < 30 ml/min/1.73m2, or history of urinary tract infection/genital yeast infection were excluded. They received oral dapagliflozin (Forxiga) 10 mg/day for 24 weeks.

The primary outcomes are the change of liver inflammation marker (serum ALT level)or fibrosis parameters after 24 weeks treatment. The adverse events were also recorded. The severity of liver fibrosis was determined using NAFLD-fibrosis score and ultrasound-based elastography method (ARFI).

Total 6 visits Visit 1 (screening): US, ARFI, body composition measurement, BP, BMI, Waist circumference, body fat (%), AST/ALT, albumin, GGT, Cr, TG, CHO, HDL/LDL, glucose ac, HbA1C, Platelet, insulin, CRP Visit 2 (2 weeks): BP, AST/ALT, Cr Visit 3 (4 weeks): BP, BMI, Waist circumference, body fat (%), AST/ALT, albumin, GGT, Cr, TG, glucose ac, HbA1C, platelet Visit 4 (3 months):BP, BMI, Waist circumference, body fat (%), AST/ALT, albumin, GGT, Cr, TG, glucose ac, HbA1C, platelet Visit 5 (6 months): US, ARFI, body composition measurement, BP, BMI, Waist circumference, body fat (%), AST/ALT, albumin, GGT, Cr, TG, CHO, HDL/LDL, glucose ac, HbA1C, Platelet, insulin, CRP Visit 6 (Month 3 off-therapy): BP, BMI, Waist circumference, body fat (%), AST/ALT, albumin, GGT, Cr, TG, CHO, HDL/LDL, glucose ac, HbA1C, Platelet Record adverse events and number of pills left in each visits

ELIGIBILITY:
Inclusion Criteria:

* MAFLD patients (hepatic steatosis plus metabolic dysfunction
* ALT elevation (>35 U/L in male and >25 U/L in female) or FIB-4 >=1.45

Exclusion Criteria:

1. diabetes history or HbA1C> 6.5
2. cancer history
3. systolic blood pressure < 100 mmHg
4. eGFR < 30 ml/min/1.73m2
5. history of urinary tract infection/genital yeast infection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-11 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of liver inflammatory marker | 24 weeks
  the change of ALT between baseline and week 24 after treatment
Change of liver fibrosis markers between baseline and week 24 after treatment | 24 weeks
  The higher NAFLD fibrosis score (NFS), the more severe liver fibrosis (no maximal or minimal levels)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided